## **PROTOCOLLO**

Efficacia di un programma di attività fisica adattata per soggetti affetti da emofilia: studio interventistico prospettico

Codice Studio: EMO-AFA

| Studio | Efficacia di un programma di attività fisica adattata per soggetti affetti da emofilia: studio interventistico prospettico |
|---|---|
| Nome e indirizzo del<br>promotore | IRCCS Istituto Ortopedico Rizzoli<br>Via di Barbiano 1/10<br>40136 Bologna |
| Responsabile dello<br>studio/PI e centro<br>Numero/Versione/Data | Dr.ssa Farella Giuseppina Mariagrazia<br>SC MEDICINA FISICA E RIABILITATIVA<br>IRCC Istituto Ortopedico Rizzoli<br>Ver. 1.0 del 14 Novembre 2023 |
| Staff di Ricerca | SC Medicina Fisica e Riabilitativa IRCCS Istituto Ortopedico Rizzoli |
| Metodologia | |
| Tipo:<br>Fondi: | No profit non previsto |

## Firma del protocollo

#### Titolo dello studio

Efficacia di un programma di attività fisica adattata per soggetti affetti da emofilia: studio interventistico prospettico.

Acronimo dello studio/Codice: EMO-AFA

Versione del Protocollo e Data: Versione 1.0 / 14 Novembre 2023

Ho letto leggi questo protocollo e accetto di condurre questo processo in conformità con le disposizioni del protocollo, le linee guida GCP e la Dichiarazione di Helsinki.

Principal Investigator

Firma, Data

Dr.ssa Farella Giuseppina Mariagrazia

Jin seffine Pariforme Forelle

01/12/2023

# **INDICE**

| LISTA DEGLI ACRONIMI | 5 |
|---------------------------------------------|----|
| 2. STATO DELL'ARTE E RAZIONALE DELLO STUDIO | 6 |
| 2.1 Introduzione | 6 |
| 2.2 Emofilia | |
| 3. OBIETTIVO DELLO STUDIO | 8 |
| 3.1 Endpoint dello Studio | 9 |
| 3.1.1 Endpoint Primario | 9 |
| 3.1.2 Endpoint secondari | 9 |
| 4. DISEGNO DELLO STUDIO | |
| 4.1 Setting dello Studio | |
| 4.2 Criteri di inclusione/esclusione | |
| 4.3 Popolazione dello studio | 11 |
| 4.4. Durata dello Studio | 11 |
| 4.5 Valutazioni | |
| 4.5.1 Valutazione basale | |
| 4.5.2 Valutazione a 3 mesi | |
| 4.5.3 Valutazione di 6 mesi | |
| 4.6 Programma di esercizio | |
| 4.7 Aderenza al programma di esercizi | |
| 4.8 Strategia per migliorare l'aderenza | |
| 4.9 Sicurezza dei partecipanti | |
| 4.10 Registrazione degli Eventi Avversi | |
| 5 ASPETTI AMMINISTRATIVI | _ |
| 5.1 Raccolta e Gestione dei Dati | |
| 5.2 Analisi Statistica | |
| 5.3 Deviazione del Protocollo | |
| 5.4 Principi Etici | |
| 5.5 Consenso Informato e Riservatezza | |
| 5.6 Confidenzialità | |
| 5.7 Report e Pubblicazione dei Risultati | |
| 5.8 Conflitto di Interessi | _ |
| 5.9 Conclusione dello studio | |
| 5.10 Archivio della documentazione | 18 |
| 5.11 Persone di riferimento | 18 |
| BIBLIOGRAFIA | 18 |

# LISTA DEGLI ACRONIMI

AE: artropatia emofilica

FISH: Functional Independence Score in Hemophilia

MD: Medical Doctor ROM: range of motion,

6MWL: il 6-minute Walking Test TSK: Tampa Scale of Kinesiophobia WFH: Word Federation of Hemophilia HJHS: Hemophilia joint health score

HAL: Questionario Hemophilia Activity List

TUG: Time Up Go

VAS: Scala Analogica Visiva

QoL: Quality of Life

STAMPA: Scienze e Tecniche dell'Attività Motoria Preventiva e Adattata

OMS: Organizzazione Mondiale della Sanità

ECA: eventi clinici avversi PI: principal investigator

# 2. STATO DELL'ARTE E RAZIONALE DELLO STUDIO

## 2.1 Introduzione

Gli studi epidemiologici confermano l'importanza dell'attività fisica per prevenire diverse malattie. L'attività fisica può prevenire l'incidenza di varie malattie, per esempio quelle cardiovascolari e va oltre alla prevenzione (1).

Nelle persone con emofilia, la condizione fisica, forza muscolare, resistenza aerobica, resistenza anaerobica e la propriocezione sono tutte diminuite. In questi soggetti aumenta il rischio di lesioni e si stabilisce un circolo vizioso difficile da spezzare: dolore, immobilità, atrofia, instabilità articolare e ripetuti episodi di sanguinamento (5). Nell'emofilia, le attività fisiche e/o attività sportive non erano raccomandate fino agli anni Settanta (per il rischio di sanguinamento in assenza di una adeguata terapia sostitutiva), quindi i pazienti emofilici non avevano la possibilità di utilizzare l'attività fisica come mezzo di prevenzione e riabilitazione. Ancora trent'anni fa, si consigliava loro di essere attivi solo quando necessario per gestire la vita quotidiana. L'inattività era considerata una forma adeguata di protezione per evitare le emorragie articolari. Ma l'inattività, tuttavia, non consente lo sviluppo di muscoli del corpo forti e ben coordinati che è una condizione preliminare per una protezione ottimale delle articolazioni. Il conseguente squilibrio muscolare combinato con disfunzioni nel movimento può portare un aumento dell'instabilità delle articolazioni che aumenta l'incidenza delle emorragie articolari e la conseguente artropatia emofiliaca (AE) (8). Negli ultimi due decenni la possibilità di effettuare la terapia sostitutiva con regolarità in regime di profilassi ha ridotto il numero di eventi emorragici e la conseguente artropatia consentendo inoltre di avviare i pazienti alla attività fisica in sicurezza.

Vi è oggi un accordo sull'importanza di attività fisiche selezionate anche per i pazienti emofilici, in modo che l'esercizio guidato da un allenatore esperto possa essere raccomandato (8).

## 2.2 Emofilia

L'Emofilia è una malattia emorragica congenita in cui il sangue non può coagulare adeguatamente a causa dell'assenza o della carenza funzionale di un fattore della coagulazione. I due tipi più comuni sono emofilia A quando il fattore carente è il fattore VIII e l'emofilia B quando il fattore carente è il IX. Si stima che l'emofilia A rappresenti l'80-85% di tutti i casi di emofilia; l'emofilia B si stima che rappresenti il 15-20% di tutti i casi di emofilia. La prevalenza stimata alla nascita è di 24,6 casi su 100.000 maschi per tutte le gravità di emofilia A (9,5 casi per l'emofilia A grave) e 5,0 casi per 100.000 maschi per tutte le gravità dell'emofilia B (1,5 casi per l'emofilia B grave) (2-3).

La malattia è trasmessa senza differenze geografiche e di popolazione come carattere recessivo legato al sesso perché codificata da geni presenti sul cromosoma X.

In base al livello di attività biologica del Fattore VIII o IX si distinguono diverse forme di Emofilia (3):

- Forma lieve caratterizzata da una riduzione del livello del fattore tra il 40% e il 5%;
- Forma moderata dove il livello del fattore è compreso tra il 5% e l'1%;
- Forma severa quando il livello del fattore è inferiore all'1% o assente.

Il sintomo principale nella persona con emofilia è il sanguinamento o emorragia. La gravità delle manifestazioni emorragiche nell'emofilia è generalmente correlata al grado di carenza del fattore di coagulazione.

Le persone con emofilia lieve possono non avere necessariamente problemi di sanguinamento fino a quando non subiscono un grave trauma o un intervento chirurgico. Le persone con emofilia grave, più comunemente, sperimentano emorragie spontanee nelle articolazioni, nei muscoli e negli organi interni. Il sanguinamento si manifesta in ugual modo sia nel tipo A sia nel tipo B (5). L'entità del sanguinamento è variabile e strettamente collegata alla gravità della malattia e alla causa meccanica scatenante.

L'emorragia più frequente è quella che avviene all'interno delle articolazioni sinoviali (emartro). La causa primaria dell'emartro è l'inefficacia del processo coagulativo, che accentua, in maniera proporzionale alla gravità dell'emofilia, ogni minima sollecitazione sul distretto: trauma o contusione, piccole distorsioni o lacerazioni di legamenti, sinovia o cartilagine. Le aree principalmente colpite sono le articolazioni di caviglie, ginocchia e gomiti. La maggior parte delle volte le emorragie articolari sono accompagnate da dolore, gonfiore, febbre e perdita di mobilità nell'articolazione in questione. Inoltre, il solo sanguinamento può causare cambiamenti strutturali e neuromuscolari nelle articolazioni colpite. Sanguinamenti ripetuti nella stessa articolazione portano alla artropatia emofilica che è una forma secondaria e infiammatoria di artrosi. Con l'avanzare dell'età della persona la frequenza degli emartri rispetto alla totalità delle emorragie cresce.

Colpendo le articolazioni, il versamento genera un processo che richiama in loco fattori dell'infiammazione. Il contatto ripetuto del sangue con le componenti articolari causa l'insorgenza di sinoviti, inizialmente acute e successivamente croniche, associate alla degenerazione della cartilagine articolare e al rimaneggiamento dell'osso subcondrale, portando all'insorgenza dell'artropatia emofilica (AE), che si caratterizza per la degenerazione di tutte le componenti articolari.

L'artropatia emofilica è considerata la malattia articolare più comune nelle persone con emofilia. Nel corso dell'artropatia emofila si verificano ulteriori adattamenti funzionali del sistema muscolo-scheletrico, come la perdita di mobilità articolare, contratture o atrofie nel sistema muscolare circostante. Questi adattamenti si traducono in limitazioni delle prestazioni fisiche. Oltre alle ridotte capacità coordinative e al deficit di forza, le persone affette da emofilia presentano un'attività fisica generalmente ridotta e una diminuzione delle prestazioni di resistenza. In particolare, le capacità motorie di forza, coordinazione e mobilità giocano un ruolo essenziale in termini di mantenimento della funzione articolare. I deficit di queste capacità motorie si traducono in un maggiore stress per l'articolazione, il che porta di nuovo a un maggiore rischio di emorragie. Emerge un circolo vizioso che consiste in un aumento delle emorragie, un declino della struttura e della funzione articolare e una riduzione delle prestazioni fisiche.

Il dolore può essere una componente invalidante importante nelle persone con AE: esso può presentarsi sia durante gli episodi emorragici acuti, sia in assenza di emorragie in atto come conseguenza della degenerazione articolare. In questo secondo caso il dolore può accompagnare la persona per la maggior parte delle attività quotidiane e indurne l'autolimitazione, con conseguenti ricadute anche sulla partecipazione sociale. Gurcay et al. (6) ha evidenziato, in giovani emofilici, una significativa riduzione del dolore dopo l'effettuazione di un programma di rinforzo isometrico e isotonico e dopo esercizi specifici per la propriocezione. Altri autori (7) hanno osservato riduzione del dolore in adulti emofilici a seguito dell'esecuzione di esercizi di rinforzo specifici per gli arti inferiori e per l'equilibrio.

Le persone con emofilia, oltre ad avere problemi al sistema muscolare, possono andare incontro a problemi al sistema scheletrico, riducendo la densità ossea (8).

Per i soggetti con problematiche muscoloscheletrica significative, è importante incoraggiare l'attività fisica contro resistenza per promuovere lo sviluppo e il mantenimento di una buona densità ossea (8).

L'attività fisica adattata aiuta non solo a rafforzare i muscoli, preservare e possibilmente migliorare la funzione articolare e il range di movimento (ROM) ma anche ad aumentare la circolazione articolare fornendo così nutrimento alla cartilagine (9-16).

L'attività fisica adattata dovrebbe essere incoraggiata per mantenere una buona forma fisica e per promuovere un normale sviluppo neuromuscolare (17-18).

L'attività fisica adattata sembra essere un modo efficace per migliorare la qualità della vita dei soggetti emofilici, con una bassa incidenza di eventi avversi correlati.

Siqueira et al. (17), evidenziano come la maggior parte degli studi presenti in letteratura mostra un'efficacia di un protocollo di esercizi sia in ambiente acquatico sia a secco, andando in particolare ad incidere sul range di movimento, forza, equilibrio e capacità aerobica.

Un programma di attività fisica adattata per soggetti emofiliaci dovrebbe focalizzarsi su (17-18):

- Forza muscolare per migliorare le reazioni dell'organismo alle variazioni di carico e incrementare l'efficacia del controllo durante i movimenti;
- Mobilità articolare e flessibilità muscolare con lo scopo di aumentare/mantenere il "range of motion" (ROM) e prevenire lesioni muscolo-articolari;
- Propriocezione ed equilibrio per mantenere un buon controllo posturale, finalizzata al mantenimento o al ripristino della corretta coordinazione senso-motoria, che può essere parzialmente compromessa a causa della riduzione di forza, del dolore o della degenerazione articolare conseguente alle ripetute emorragie
- Attività aerobica per migliorare/mantenere la funzione cardio/vascolare dell'organismo.

Per le persone con emofilia, la World Federation of Hemophilia (WFH) raccomanda la promozione dell'attività fisica regolare, con particolare attenzione al mantenimento della salute delle ossa, rafforzamento muscolare, coordinazione, funzionamento fisico, peso corporeo sano e autostima positiva.

La rilevanza delle problematiche muscolo-scheletriche correlate a questa patologia e le relative conseguenze sul piano funzionale e della partecipazione alla vita sociale, rendono necessaria, quindi, una presa in carico globale delle persone affette da emofilia. Questo richiede piani di valutazione e trattamenti personalizzati e specifici, in modo tale da rispondere alle diverse e specifiche necessità di ciascun paziente.

Il paziente emofilico dovrebbe essere seguito da un team multidisciplinare di professionisti comprendente fra gli altri un esperto in malattie della coagulazione, un medico fisiatra, un laureato in fisioterapia (8) e un laureato magistrale in scienze e tecnica dell'attività motoria preventiva e adattata.

Questo studio apporterà maggiori conoscenze a livello quali-quantitativo del beneficio che l'attività fisica può portare alle persone con emofilia in linea con le Linee Guida della OMS che promuovono l'attività fisica a qualsiasi età e a qualsiasi tipo di abilità.

# 3. OBIETTIVO DELLO STUDIO

Il presente studio ha come obiettivo di valutare la modificazione della capacità funzionale indotta da un programma di attività fisica adattato in soggetti con emofilia.

## 3.1 Endpoint dello Studio

## 3.1.1 Endpoint Primario

L'endpoint primario è la variazione della capacità funzionale calcolata come differenza tra la valutazione basale e la valutazione a 3 e a 6 mesi del 6 Minutes Walking Test misurato con il G-Walk (BTS Bioengineering S.p.A).

## 3.1.2 Endpoint secondari

Gli endpoint secondari includeranno la valutazione basale e a 3 e a 6 mesi della qualità della vita e di alcuni domini che influenzano la qualità della vita

I questionari e i test utilizzati sono tutti validati e saranno:

Functional Independence Score in Hemophilia (FISH) (19) è un questionario che viene effettuato da un operatore per valutare l'autonomia nello svolgimento di otto attività della vita quotidiana: igiene personale, mangiare, vestirsi, compiere trasferimenti dalla sedia, accovacciarsi, camminare, salire le scale, correre. Ogni attività è misurata in funzione della quantità di assistenza necessaria per eseguirla.

- Hemophilia joint health score (HJHS) (20) è una scala compilata da un operatore per la valutazione dello stato di salute delle articolazioni. La scala HJHS misura la salute articolare nei domini della struttura del corpo e della funzione (biomeccanica) delle strutture più frequentemente colpite da emorragia in pazienti affetti da emofilia: le ginocchia, le caviglie e i gomiti.
- Tampa Scale of Kinesiophobia (TSK) (21) è un questionario compilato dal paziente per valutare la paura del movimento. Questa scala è parametro di valutazione internazionale con il quale si è evidenziata una persistente e costante preoccupazione del tutto ingiustificata nel dover compiere movimenti per paura di procurarsi dolore o danni, capace di compromettere tutte le azioni di vita quotidiana anche lavorative con chiare ripercussioni anche di carattere socio-economico.
- Questionario Hemophilia Activity List (HAL) (22) è un questionario compilato dal paziente sulle limitazioni delle attività. La scala HAL misura l'impatto dell'emofilia sulle capacità funzionali nel soggetto adulto. È composta da 42 domande che indagano 7 domini: 1. Sdraiato / Seduto / In ginocchio / In piedi, 2. Funzioni delle gambe, 3. Funzioni delle braccia, 4. Trasporti, 5. Cura personale, 6. Attività domestiche, 7. Attività di svago e sportive.
- Forza Muscolare (test eseguito da operatore) tramite
  - 30" Chair stand test (23)
  - Arm curl test (28)
  - Massima forza isometrica dei flessori ed estensori dell'anca tramite Hand held; (24)
  - Massima forza isometrica dei flessori ed estensori del ginocchio tramite hand held (24)
- Equilibrio (test eseguito da operatore)
  - Single leg stand test (25)

- Time Up Go (TUG) (26)
- Scala Analogica Visiva (VAS) nelle articolazioni bersaglio (27) compilata dal paziente.

L'aderenza di ciascun paziente al programma di esercizi verrà monitorata. L'aderenza verrà misurata come percentuale di sessioni di allenamento effettivamente eseguite / numero totale di sessioni di allenamento programmate.

Nel contesto della valutazione dell'adesione al programma, la soddisfazione dei partecipanti al programma di attività fisica sarà effettuato a 3-6 mesi con un questionario specifico basato sulla scala Likert e le ragioni per abbandonare il programma di esercizi (28) (domande con risposte strutturate, compilato dal paziente).

# 4. DISEGNO DELLO STUDIO

Studio clinico interventistico.

# 4.1 Setting dello Studio

I pazienti affetti da emofilia A o B saranno reclutati presso l'ambulatorio MEC fisio della SC Medicina Fisica e Riabilitativa dell'Istituto Ortopedico Rizzoli, dedicato all'attività di consulenza fisiatrica per i pazienti affetti da emofilia in carico alla SSD Malattie Emorragiche Congenite dell'IRCCS Azienda Ospedaliero-Universitaria di Bologna che continuerà a seguirli per il monitoraggio ematologico come da pratica clinica. La partecipazione sarà proposta ai soggetti che afferiscono per visite di controllo e che rientrano nei criteri di inclusione.

Inoltre, per facilitare il reclutamento dei soggetti, lo studio sarà pubblicizzato tramite comunicazione alle associazioni e federazioni dei soggetti emofilici.

Se idoneo allo studio, al soggetto sarà richiesto di firmare il consenso informato e i dati personali (nome e cognome, indirizzo, numero di telefono) saranno registrati solo sul modulo di consenso informato con il codice dello studio. In tutti gli altri format utilizzati nello studio, i partecipanti saranno identificati con un codice univoco di studio.

Durante lo studio, a tutti i pazienti sarà raccomandato di mantenere la terapia farmacologica, come da indicazione del medico.

Tutti i soggetti reclutati saranno valutati al baseline, a 3 mesi e a 6 mesi dal personale di ricerca. Tutte le valutazioni mediche e gli score funzionali saranno effettuati presso l'ambulatorio dedicato della struttura Complessa Medicina Fisica e Riabilitativa dell'Istituto Ortopedico Rizzoli.

I questionari e gli score funzionali saranno eseguiti dal personale universitario afferente al Dipartimento di Scienze di Qualità della vita dell'Università di Bologna presso la palestra del Centro sportivo Record che sarà anche la sede della attività fisica adattata.

## 4.2 Criteri di inclusione/esclusione

#### Criteri di inclusione

- Diagnosi di emofilia A o B;
- Firma del consenso informato;
- Disponibilità di un certificato medico per attività non agonistica
- Ambo i sessi con età compresa tra 18 anni e 80 anni.

#### Criteri di esclusione

- Sanguinamenti in atto
- Gravi deformità articolari che impediscano l'esercizio
- Insufficienza delle funzioni comunicative e / o sensoriali così gravi da rendere impossibile la comprensione o l'esecuzione delle istruzioni del formatore (demenza, afasia, cecità, sordità)
- Insufficienza cardiaca (classe NYHA> 2)
- Angina instabile
- Malattia polmonare che richiede ossigenoterapia
- Arteriopatia periferica sintomatica
- Infarto del miocardio o ricovero ospedaliero nei 6 mesi precedenti
- Ipotensione ortostatica sintomatica
- Ipertensione in scarso controllo farmacologico (diastolica> 95 mmHg, sistolica> 160 mmHg)
- Rilevanti condizioni neurologiche che compromettono la funzione motoria o cognitiva
- Qualsiasi altra condizione che i medici della SC di Medicina Fisica e Riabilitativa e SSD Malattie Emorragiche Congenite ritenga controindicata per la partecipazione a un programma di esercizi di lieve/moderata intensità.

## 4.3 Popolazione dello studio

La dimensione del campione è stata calcolata attraverso una power analysis a priori basata sull'outcome primario dello studio, ovvero la distanza percorsa nel 6 Minute Walking Test (6MWT), valutato prima dell'intervento con protocollo di attività fisica e ad un follow up di 6 mesi. È stato considerato come riferimento un recente studio pilota interventistico presente in letteratura con razionale simile (18). A partire da tale studio, nel quale è stato utilizzato il 6MWT con valutazione nell'immediato post-intervento e a 6 mesi di follow-up, sono stati riportati una deviazione standard pari a 21.1m per il follow-up e 18.8 m per il baseline e differenza tra le medie baseline e a 6 mesi di 23.9 m. Da questo, è stato ricavato un effect size pari 1.19 (considerato "elevato"). Allo scopo di mantenere una valutazione campionaria più conservativa, per questo studio viene ipotizzato un effect size minore di quello ricavato da letteratura, pari a 0.8. La power analysis è quindi stata effettuata utilizzando un t-test a una coda per dati appaiati con un errore  $\alpha$ =0.05 e un sample power (1- $\beta$ ) di 0.8, risultando in un numero minimo di 12 pazienti, in linea con la letteratura corrente. È stata quindi considerata una percentuale di drop-out del 25%. La dimensione campionaria minima viene quindi stimata in 16 pazienti.

## 4.4. Durata dello Studio

Il periodo di intervento dell'attività fisica per ciascun partecipante allo studio durerà 6 mesi.

Il progetto avrà una durata totale di 14 mesi suddivisi come segue:

- Mesi 1-6 Selezione, arruolamento e valutazione basale dei pazienti
- Mesi 1-12 Attività fisica
- Mesi 12-14 Analisi dei dati

L'approvazione del Comitato Etico sarà considerata come la data di inizio della sperimentazione.

## 4.5 Valutazioni

#### 4.5.1 Valutazione basale

I dati sono registrati dal personale clinico e di ricerca in un modulo specifico di valutazione basale.

Lo staff di ricerca raccoglie informazioni sulle caratteristiche generali (essenziali per contattare i pazienti e per fornire informazioni su fattori che possono influenzare l'aderenza al programma di esercizi), capacità funzionale, forza muscolare, mobilità articolare, funzione motoria, stile di vita, salute e qualità della vita (QoL).

Al fine di promuovere la coerenza nella qualità dei dati, tutti i valutatori saranno sottoposti a un corso di formazione sulla gestione degli strumenti di valutazione dello studio. Ai formatori viene inoltre fornito un manuale che fornisce istruzioni chiare su come amministrare gli strumenti di valutazione.

Saranno valutati i seguenti domini:

- Dati generali
- Capacità funzionale
- Oualità della vita
- Funzione motoria

#### 4.5.2 Valutazione a 3 mesi

A 3 mesi vengono ripetute le misure quali:

- Capacità funzionale
- Funzione motoria

Inoltre, a tutti i partecipanti verrà chiesto di compilare un questionario strutturato in merito a:

- Opinione sul programma di esercizi cui hanno partecipato [risposte strutturate basate su una scala Likert];
- I motivi principali per cui hanno abbandonato il programma di esercizi [domanda con risposte strutturate].

#### 4.5.3 Valutazione di 6 mesi

Vengono ripetute le misure tutti effettuate alla baseline, quindi sui seguenti domini:

- Capacità funzionale;
- Qualità della vita;
- Funzione motoria.

Inoltre, a tutti i partecipanti verrà chiesto di compilare un questionario strutturato in merito a:

- Opinione sul programma di esercizi cui hanno partecipato [risposte strutturate basate su una scala Likert];
- I motivi principali per cui hanno abbandonato il programma di esercizi [domanda con risposte strutturate].

# 4.6 Programma di esercizio

Il programma di esercizi utilizzato ha lo scopo di migliorare la mobilità articolare, la forza muscolare, l'equilibrio statico e dinamico, la coordinazione motoria.

Il programma è strutturato in sessioni di 1 ora di 2 giorni / settimana e dura 6 mesi.

Ogni sessione è strutturata nelle seguenti sezioni: riscaldamento, parte centrale (dove saranno inseriti esercizi di forza, di equilibrio, di coordinazione), defaticamento.

Il trainer adotterà il programma di esercizi alle esigenze e alle preferenze dei partecipanti.

#### Il protocollo definisce:

- Strategie per istruire i pazienti e verificare la corretta e sicura esecuzione dei compiti motori
- Criteri per l'avanzamento del carico di lavoro e il numero di ripetizioni per adattarsi a ogni singola capacità funzionale

L'attività fisica verrà eseguita in spazi/palestre, che hanno stipulato accordi formali con l'Università di Bologna o all'interno dei locali delle associazioni oppure online sempre sotto la diretta supervisione di un trainer laureato magistrale in Scienze e Tecniche delle attività motoria preventive e adattate (STAMPA).

#### Altre attività consigliate

Ai soggetti verrà richiesto di eseguire per altri 2/3 giorni della settimana una delle seguenti attività: camminata veloce, ciclismo o nuoto. La durata raccomandata di queste attività sarà di 20-40 minuti. In questo modo, i pazienti raggiungeranno la quantità di esercizio alla settimana di 150 minuti raccomandata dall'OMS (http://www.who.int/dietphysicalactivity/factsheet\_olderadults/en/). I pazienti sono tenuti a registrare anche l'esecuzione di queste attività in un diario.

# 4.7 Aderenza al programma di esercizi

#### Procedura per monitorare l'aderenza

Per ciascun partecipante, la partecipazione al programma di esercizi verrà registrata dal trainer in un registro all'inizio di ogni sessione di ginnastica.

Ai partecipanti verrà inoltre richiesto di registrare le "attività aggiuntive" in un diario.

L'aderenza verrà stimata come percentuale delle sessioni effettivamente eseguite rispetto al numero totale teorico di sessioni.

## 4.8 Strategia per migliorare l'aderenza

Se un partecipante perde una o due sessioni consecutive ne viene chiesto il motivo alla prima sessione di allenamento a cui partecipa. Se un partecipante perde tre sessioni consecutive il trainer lo contatterà telefonicamente per chiedere la motivazione dell'assenza e incoraggiare l'aderenza, se del caso. Il trainer registra la data dell'assenza e la motivazione nel registro del paziente.

# 4.9 Sicurezza dei partecipanti

Data la persistenza della pandemia di COVID-19, tutte le attività dello studio riguardanti sia le valutazioni che le attività in palestra dei partecipanti e dei ricercatori saranno svolte secondo le disposizioni dell'ultimo Decreto del Presidente del Consiglio dei Ministri e dei relativi aggiornamenti e le linee guida definite dall'Ufficio per lo Sport della Presidenza del Consiglio dei Ministri.

I danni dovuti all'esercizio fisico sono raramente riportati nella letteratura pubblicata e generalmente includono lesioni muscolo-scheletriche minori. Pertanto esiste ora un considerevole corpo di dati che dimostrano la sicurezza di iniziare l'esercizio fisico in questi contesti in coorti con comorbidità multiple e preesistente compromissione funzionale e disabilità. Nonostante ciò, la sicurezza dei partecipanti rimane una delle principali preoccupazioni in questo studio e un comportamento prudente è stato adottato per affrontare gli eventi clinici (ECA)

Gli eventi avversi derivati dall'esecuzione dell'esercizio fisico sono raramente riportati nella letteratura pubblicata e generalmente includono lesioni muscoloscheletriche minori.

Pertanto, esiste ora un considerevole corpus di dati per dimostrare la sicurezza di iniziare l'esercizio in questi contesti in coorti con comorbilità multiple e disabilità e disabilità funzionali preesistenti.

Ciononostante, la sicurezza dei partecipanti rimane una delle maggiori preoccupazioni in questo studio ed è stato adottato un comportamento cautelativo per far fronte agli eventi clinici avversi (ACE).

#### Ruolo del trainer

L'intensità dell'esercizio non deve superare quanto indicato, adattando il ritmo alla capacità del singolo soggetto. Durante le sessioni iniziali il trainer propone precauzioni da prendere nella vita di tutti i giorni (sdraiarsi e alzarsi da terra e dal letto, alzarsi / sdraiarsi sul letto, allacciarsi le scarpe, raccogliere oggetti da terra, ecc.);

## Numero di partecipanti per gruppo

Per poter avere un miglior monitoraggio dei soggetti e per motivi di sicurezza il numero massimo di partecipanti in ciascuna sessione non deve superare le 5 unità.

#### Gestione degli eventi clinici avversi (ECA)

In caso di eventi avversi catastrofici (ad esempio cadute traumatiche), se necessario, è compito del trainer attivare le procedure di intervento dei servizi di emergenza comunitari (118). Il PI dello studio svolge un'indagine e prende le precauzioni necessarie per evitare che l'evento si ripeta. Se la causa è considerata il programma di esercizi, quest'ultimo può essere modificato. Durante ogni sessione il trainer informa di eventuali cambiamenti nello stato di salute dei partecipanti durante e al di fuori del programma di esercizi (ad esempio l'insorgenza di dolori articolari o muscolari).

#### Ruolo del medico di Medicina di Base e del Medico Specialista di riferimento

Il medico di famiglia è informato per lettera dell'inclusione del paziente nel progetto di studio. Se durante lo studio si verifica qualsiasi evento menzionato nel paragrafo "Criteri di esclusione", il medico di medicina di Base comunicherà l'evento al PI dello studio che procederà a una rivalutazione dei criteri di inclusione/esclusione nello studio e alla eventuale revoca del consenso. Di conseguenza il paziente verrà escluso dallo studio e le motivazioni verranno registrate.

## 4.10 Registrazione degli Eventi Avversi

Gli eventi clinici avversi (ECA) che si verificheranno per i partecipanti saranno accuratamente registrati nei registri durante tutto lo studio. Per ogni soggetto verranno registrati gli eventi clinici avversi durante le sessioni di allenamento e al di fuori di essi.

Gli eventi clinici avversi saranno registrati dai trainer in ogni sessione di allenamento. Nel caso di 3 assenze consecutive, il trainer contatterà telefonicamente il paziente per verificare se la causa della mancata partecipazione alle sessioni in palestra fosse dovuto ad evento clinico avverso.

Sulla base dei registri, un ECA è classificato:

- 1) Per gravità come:
  - a. Grave: se l'evento clinico avverso ha comportato un ricovero / accesso al pronto soccorso
- b. Moderato: se l'evento clinico avverso ha richiesto l'intervento di un medico e / o la modifica della normale terapia farmacologica
- c. Lieve: se l'evento clinico avverso non ha richiesto l'intervento medico e / o la modifica della normale terapia farmacologica
- 2) Per il luogo in cui si è verificato l'evento:
  - a. casa
  - b. fuori casa
  - c. In palestra
- 3) A seconda dell'apparato / sistema interessato.

# **5 ASPETTI AMMINISTRATIVI**

## 5.1 Raccolta e Gestione dei Dati

I dati clinici richiesti dal protocollo verranno raccolti in forma pseudonimizzata dal personale designato dal PI in una Scheda Raccolta Dati (CRF) elettronica.

Tutti i moduli cartacei saranno verificati e archiviati in armadietti bloccati. I dati dello studio registrati nella visita di reclutamento del paziente saranno inseriti direttamente nel database CRF accessibile tramite password solo dal personale designato dal PI. I dati derivati dai questionari e dagli score funzionali saranno registrati su moduli cartacei e saranno successivamente inseriti in

CRFp. Il materiale cartaceo sarà quindi archiviato in armadietti bloccati presso la SC Medicina Fisica E Riabilitativa.

. Il database verrà chiuso una volta dichiarato completo e accurato. Eventuali modifiche ai dati dopo la chiusura possono essere eseguite dal personale proposto solo quando si inseriscono i dati con il consenso preventivo del PI.

Il PI è assistito, nell'ambito dello studio, dallo staff di ricerca per la gestione, l'analisi e l'interpretazione dei dati.

#### 5.2 Analisi Statistica

Le variabili qualitative saranno riassunte in termini di frequenza, quelle quantitative in termini di deviazione media e standard per gruppo e per i tre tempi di valutazione. Per l'analisi dei risultati verrà utilizzato il principio dell'intenzione di trattare, adattandosi all'adesione al programma di esercizi. Sarà effettuato il confronto fra i dati al basale e quelli rilevati a 3 e a 6 mesi: per l'analisi sarà utilizzato il test di Friedman.

## 5.3 Deviazione del Protocollo

Lo studio deve essere condotto come descritto nel presente protocollo. Il PI non implementerà alcuna deviazione o modifica del protocollo senza una revisione preventiva e l'approvazione documentata dell'emendamento da parte del Comitato Etico, salvo ove necessario per eliminare un rischio immediato (i) per studiare le materie.

- a. Deviazioni del protocollo
  - Eventuali non aderenze al protocollo di studio che non comportano criteri di inclusione / esclusione, criteri di variabili oggettive primarie e / o linee guida di buona pratica clinica saranno considerate minori e non incidono sullo studio;
- b. Violazioni del protocollo
  - Qualsiasi violazione del protocollo comporterà una significativa divergenza rispetto al protocollo, vale a dire la non aderenza da parte del paziente o dello sperimentatore ai criteri di inclusione / esclusione specifici del protocollo, criteri delle variabili dell'obiettivo primario e / o linee guida GCP. Tutti gli investigatori saranno responsabili di comunicare al PI qualsiasi violazione del protocollo osservata entro 24 ore. Il PI deciderà se il paziente può continuare nello studio o se deve essere ritirato da esso.
- c. Eccezioni del protocollo
  - Per motivi di politica, il PI non concede eccezioni ai criteri di ingresso specifici del protocollo per consentire ai pazienti di accedere a uno studio. Se in circostanze straordinarie tale azione è considerata eticamente, dal punto di vista medico o scientificamente giustificata per un particolare paziente, prima che al paziente sia permesso di entrare nello studio sarà richiesta la previa approvazione scritta del PI.

# 5.4 Principi Etici

Il protocollo di ricerca e i relativi documenti saranno inviati prima di iniziare lo studio alle autorità competenti e al comitato etico per la sua approvazione. Lo sperimentatore responsabile assicurerà che lo studio venga condotto in accordo alla Dichiarazione Helsinki nella sua versione più aggiornata (Fortaleza, Ottobre 2013), nonché con tutta la normativa nazionale ed internazionale applicabile alla ricerca clinica.

Il protocollo è stato scritto e lo studio sarà condotto secondo i principi delle ICH-GCP.

## 5.5 Consenso Informato e Riservatezza

Tutti i pazienti saranno informati degli obiettivi dello studio e dei possibili rischi e benefici che deriveranno dalla partecipazione allo studio. L'investigatore informerà chiaramente che il paziente è libero di rifiutare la partecipazione allo studio e che può revocare il consenso in qualsiasi momento e per qualsiasi motivo e che la partecipazione non ha alcun costo per il soggetto stesso. I soggetti saranno informati della massima riservatezza dei dati dello studio e che i medesimi dati potranno essere rivisti a fini di prova solo da persone autorizzate I medici della SC di Medicina Fisica e Riabilitativa dell'Istituto Ortopedico Rizzoli avranno l'incarico di acquisire il consenso informato e il consenso al trattamento dei dati dai pazienti presso la medesima SC.

Per partecipare allo studio ogni paziente dovrà fornire il consenso informato scritto nonché il consenso al trattamento dei suoi dati personali.

Il modulo di consenso informato scritto sarà firmato e datato personalmente dai pazienti. L'investigatore firmerà anche il modulo di consenso informato e manterrà l'originale sul sito e consegnerà al paziente una copia dell'originale.

I dati sensibili verranno trattati secondo la normativa vigente dal responsabile dello studio. Inoltre, i partecipanti potranno ritirare in ogni momento il consenso alla partecipazione, senza alcuna conseguenza.

La tutela delle informazioni personali fornite dai soggetti avverrà secondo la normativa vigente in materia di protezione dei dati personali. In linea con la normativa internazionale riguardo la protezione dei dati, verranno adottate le seguenti misure:

Il materiale cartaceo verrà conservato in armadi dedicati chiusi a chiave e non accessibili a soggetti non autorizzati;

## 5.6 Confidenzialità

Tutti i pazienti inclusi nello studio saranno identificati con un codice numerico, in modo che i dati personali saranno resi pseudoanonimi e utilizzati nel rispetto della normativa in vigore in materia di privacy. I dati verranno conservati dallo sperimentatore per il tempo necessario alla produzione scientifica.

Al fine di garantire la riservatezza dei dati delle sperimentazioni cliniche come disposto dalla normativa nazionale ed europea applicabile, i dati saranno accessibili solo al promotore dello studio e i suoi designati, per le procedure di monitoraggio/auditing, allo sperimentatore e i collaboratori, e al Comitato etico del centro in cui viene condotta la ricerca e alle autorità sanitarie preposte.

Lo sperimentatore e l'Istituto consentiranno l'accesso ai dati e alla documentazione di origine per il monitoraggio, l'audit, la revisione del Comitato etico e le ispezioni dell'Autorità sanitaria, ma conservando riservatezza dei dati personali in accordo alla normativa vigente.

## 5.7 Report e Pubblicazione dei Risultati

Lo sperimentatore principale si impegna a produrre il report finale, pubblicare tutti i dati raccolti come descritto nel protocollo e garantire che i dati siano riportati responsabilmente e coerentemente.

In particolare, la pubblicazione dei dati derivanti dal presente studio avverrà indipendentemente dai risultati ottenuti.

La trasmissione o diffusione dei dati, per il tramite di pubblicazioni scientifiche e/o di presentazione a congressi, convegni e seminari, avverrà esclusivamente a seguito dell'elaborazione meramente statistica degli stessi, o comunque in forma assolutamente anonima.

## 5.8 Conflitto di Interessi

Non ci sono situazioni di conflitto di interessi dei professionisti che partecipano allo studio.

#### 5.9 Conclusione dello studio

Lo Sperimentatore si impegna a comunicare l'avvenuta conclusione dello studio e ad inviare almeno un abstract o pubblicazione derivato dallo studio a chi di competenza.

## 5.10 Archivio della documentazione

Il PI è responsabile dell'archiviazione e conservazione dei documenti essenziali dello studio, prima, durante la conduzione e dopo il completamento o l'interruzione dello studio stesso, in accordo a quanto previsto dalla normativa vigente e dalle GCP e relative tempistiche.

I dati raccolti nella CRF saranno in forma rigorosamente pseudonima ed il soggetto verrà unicamente identificato con un numero/codice.

Lo Sperimentatore dovrà conservare i dati originali del paziente ed il consenso informato scritto firmato in luogo sicuro, per assicurare il mantenimento della confidenzialità e riservatezza.

## 5.11 Persone di riferimento

I numeri di telefono e le email delle persone di riferimento per la conduzione dello studio sono riportati nell'Investigator Folder presso il centro.

# **BIBLIOGRAFIA**

- World Health Organization. Global action plan on physical activity 2018-2030: more active people for a healthier world. 2018. http://apps.who.int/iris/bitstream/handle/10665/272722/9789241514187-eng.pdf
- 2. Iorio A , Stonebraker JS , Chambost H , et al. Establishing the prevalence and prevalence at birth of hemophilia in males: a metaanalytic approach using national registries . Ann Intern Med. 2019; 171 (8): 540 546;
- 3. WFH Guidelines for the Management of Hemophilia, 3rd edition Haemophilia. 2020;26(Suppl 6):1–158.
- 4. Lee CA, Berntorp EE, Keith Hoots W; Textbook of Hemophilia 3th Edition 2014 Wiley Ed;

- 5. Clausen N, Petrini P, Claeyssens-Donadel S, Gouw SC, Liesner R Similar bleeding phenotype in young children with haemophilia A and B: a cohort study. PedNet and Research of Determinants of Inhibitor development (RODIN) Study Group Haemophilia 2014; 20(6) 747–55; 5. Gurcay E, Eksioglu E, Ezer U, Cakir B, Cakci A. A prospective series of musculoskeletal system rehabilitation of arthropathic joints in young male hemophilic patients. Rheumatol Int. 2008 Apr;28(6):541-5. Epub 2007 Oct 18
- 6. Hill K, Fearn M, Williams S, Mudge L, Walsh C, McCarthy P, Walsh M, Street A. Effectiveness of a balance training home exercise programme for adults with haemophilia: a pilot study. Haemophilia. 2010 Jan;16(1):162-9;
- 7. Srivastava A, Brewer AK, Mauser-Bunschoten EP, Key NS, Kitchen S, Llinas A, Ludlam CA, Mahlangu JN, Mulder K, Poon MC, Street A; Treatment Guidelines Working Group on Behalf of The World Federation Of Hemophilia. Guidelines for the management of hemophilia. Haemophilia. 2013 Jan;19(1):e1-47;
- 8. Nied RJ, Franklin B. Promoting and prescribing exercise for the elderly. Am FamPhysician 2002; 65: 419–26.
- 9. Bennell KL, Hinman RS, Metcalf BR et al. Efficacy of physiotherapy management of knee joint osteoarthritis: a randomised, double blind, placebo controlled trial. Ann Rheum Dis 2005; 64: 906–12;
- 10. Mulvany R, Zucker-Levin AR, Jeng M et al. Effects of a 6-week, individualized, super-vised exercise program for people with bleeding disorders and hemophilic arthritis. Phys Ther 2010; 90: 509–26
- 11. Gomis M, Querol F, Gallach JE, Gonzale LM, Aznar JA. Exercise and sport in the treatment of haemophilic patients: a systematic review. Haemophilia 2009; 15: 43–54
- 12. Ettinger WH Jr, Burns R, Messier SP et al. A randomized trial comparing aerobic exercise and resistance exercise with a health education program in older adults with knee osteoarthritis. The Fitness Arthritis and Seniors Trial (FAST). JAMA 1997; 277: 25–31.
- 13. Roddy E, Zhang W, Doherty M. Aerobic walking or strengthening exercise for osteoarthritis of the knee? A systematic review. Ann Rheum Dis 2005; 64: 544–8.
- 14. Fransen M, McConnell S, Bell M. Therapeutic exercise for people with osteoarthritis of the hip or knee. A systematic review. J Rheumatol 2002; 29: 1737–45;
- 15. Fransen M, McConnell S, Hernandez-Molina G, Reichenbach S. Exercise for osteoarthritis of the hip. Cochrane Database of SystRev 2009; CD007912
- 16. Linee guida della World Federation of Hemophilia 2nd Edition
- 17. Thais Cristina Siqueira, Fábio Hech Dominski, Alexandro Andrade. Effects of exercise in people with haemophilia: An umbrella review of systematic reviews and meta-analyses. Haemophilia. 2019;25:928–937
- 18. 1Volkan Deniz, Nevin Atalay Guzel, Sébastien Lobet, Ali Bülent Antmen, Hatice Igen Sasmaz, Abdullah Kilci, Omer Cumhur Boyraz, Ozgür Gunaştı, Sanli Sadi Kurdak, Effects of a supervised therapeutic exercise program on musculoskeletal health and gait in patients with haemophilia: A pilot study. "Haemophilia" (2021)

- Poonnoose, P. M., Manigandan, C., Thomas, R., Shyamkumar, N. K., Kavitha, M. L., Bhattacharji, S., & Srivastava, A. (2005). Functional Independence Score in Haemophilia: a new performance-based instrument to measure disability. Haemophilia: the official journal of the World Federation of Hemophilia, 11(6), 598–602. <a href="mailto:μhttps://doi.org/10.1111/j.1365-2516.2005.01142.x">μhttps://doi.org/10.1111/j.1365-2516.2005.01142.x</a> §
- 20. Ribeiro, T., Abad, A., & Feldman, B. M. (2019). Developing a new scoring scheme for the Hemophilia Joint Health Score 2.1. Research and practice in thrombosis and haemostasis, 3(3), 405–411. <a href="mailto:uhttps://doi.org/10.1002/rth2.12212"><u>uhttps://doi.org/10.1002/rth2.12212</u></a>§
- 21. Monticone, Marco MD\*; Giorgi, Ines Psy†; Baiardi, Paola PhD‡; Barbieri, Massimo MD§; Rocca, Barbara Psy\*; Bonezzi, Cesare MD§ Development of the Italian Version of the Tampa Scale of Kinesiophobia (TSK-I): Cross-Cultural Adaptation, Factor Analysis, Reliability, and Validity, Spine: May 20, 2010 Volume 35 Issue 12 p 1241-1246 doi: 10.1097/BRS.0b013e3181bfcbf6
- 22. Van Genderen, F.R., Westers, P., Heijnen, L., De Kleijn, P., Van Den Berg, H.M., Helders, P.J.M. And Van Meeteren, N.L.U. (2006), Measuring patients' perceptions on their functional abilities: validation of the Haemophilia Activities List. Haemophilia, 12: 36-46. https://doi.org/10.1111/j.1365-2516.2006.01186.x
- 23. Benton, M. J., & Alexander, J. L. (2009). Validation of functional fitness tests as surrogates for strength measurement in frail, older adults with chronic obstructive pulmonary disease. American journal of physical medicine & rehabilitation, 88(7), 579–590. <a href="https://doi.org/10.1097/PHM.0b013e3181aa2ff8">https://doi.org/10.1097/PHM.0b013e3181aa2ff8</a>
- 24. Hébert, Luc J. PT, PhD; Maltais, Désirée B. PT, PhD; Lepage, Céline PT, MSc; Saulnier, Joanne PT; Crête, Mélanie PT; Perron, Marc PT, MSc Isometric Muscle Strength in Youth Assessed by Hand-held Dynamometry, Pediatric Physical Therapy: Fall 2011 Volume 23 Issue 3 p 289-299 doi: 10.1097/PEP.0b013e318227ccff
- 25. Hunt, M.A., McManus, F.J., Hinman, R.S. and Bennell, K.L. (2010), Predictors of single-leg standing balance in individuals with medial knee osteoarthritis. Arthritis Care Res, 62: 496-500. https://doi.org/10.1002/acr.20046
- 26. Podsiadlo, D. and Richardson, S. (1991), The Timed "Up & Go": A Test of Basic Functional Mobility for Frail Elderly Persons. Journal of the American Geriatrics Society, 39: 142-148. https://doi.org/10.1111/j.1532-5415.1991.tb01616.x
- 27. Boonstra, A. M., Schiphorst Preuper, H. R., Reneman, M. F., Posthumus, J. B., & Stewart, R. E. (2008). Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. International journal of rehabilitation research. Internationale Zeitschrift für Rehabilitationsforschung. Revue internationale de recherches de readaptation, 31(2), 165–169. https://doi.org/10.1097/MRR.0b013e3282fc0f93
- 28. Louangrath, Paul. (2018). Reliability and Validity of Survey Scales. 10.5281/zenodo.1322695.